CLINICAL TRIAL: NCT00277446
Title: Dietary Supplementation With Soy Isoflavones in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Lewis Smith/Professor of Medicine, Northwestern University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0456-035
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Results first posted 2011-02-24 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Asthma
Keywords: Asthma; Soy isoflavones; Eosinophils; Exhaled nitric oxide
MeSH Terms: conditions — Asthma | interventions — Soybean Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Soy isoflavones

SUMMARY:
An epidemiologic study of patients with asthma has shown that increased intake of soy isoflavones correlates with less severe asthma. In experimental animals, treatment with the soy isoflavone genistein reduces airways inflammation and hyper-responsiveness. In vitro studies performed by us have shows that genistein reduces release of inflammatory compounds by human blood eosinophils. The purpose of this pilot study is to determine whether dietary supplementation with soy isoflavones has effects in patients with asthma. 20 patients with asthma will supplement their diet with a soy isoflavone capsule for 4 weeks. Before and after the supplementation period, we will measure lung function, exhaled nitric oxide (a marker for airway inflammation), collect exhaled breath condensate to measure levels of inflammatory mediators in the airways, and isolate peripheral blood eosinophils to assess the impact of soy isoflavones on their function. We hypothesize that dietary supplementation with soy isoflavones will reduce exhaled nitric oxide level, reduce the inflammatory mediators in the exhaled breath condensate, and reduce the ability of eosinophils to release inflammatory molecules. Identifying if these hypothesized effects of soy isoflavones exist in asthma will provide a justification for further clinical studies.

DETAILED DESCRIPTION:
This is a prospective pilot study to be conducted in 20 subjects with asthma. The participant will undergo the following procedures:

1. Completion of a questionnaire that asks for information about asthma including symptoms, medications, and ability to participate in activities.
2. Measurement of exhaled nitric oxide (NO) in which subjects will breathe slowly into a tube. This test takes about 5 minutes.
3. Collection of the air exhaled from the lungs and condensing it into a liquid form. This is called an exhaled breath condensate. This procedure involves breathing slowing into a tube for a period of 15 minutes. The measurements determined by this method are exclusively for research purposes and not used in routine clinical settings.
4. Measurement of lung function with a spirometer. This involves breathing in and out forcefully through a mouthpiece.
5. Collection of 60 ml (4 tablespoons) of blood to measure genistein (the major component of the soy isoflavone) levels and eosinophil function. These measurements are also for research purposes and not routinely used clinically.

Each of the above measurements will be made before and after the 4 week period of dietary supplementation with soy isoflavones.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-50, males and females
* Physician diagnosis of asthma; requires daily asthma medication
* Moderate persistent disease (NAEPP guidelines)
* FEV1 65 to 90% of predicted
* At least 12% increase in FEV1 15-30 minutes after inhaling 2-4 puffs of albuterol or positive methacholine challenge (20% fall in FEV1 at less than 8 mg/ml) - either of these can available from the previous 2 years
* Generally good health

Exclusion Criteria:

* Oral corticosteroid use within the past 3 months
* Use of high dose inhaled corticosteroids (greater than 500 mcg of fluticasone per day or greater)
* Current or former smoker (quit less than 6 months prior to study enrollment or greater than 10 pack years)
* Recent asthma exacerbation (within 6 weeks)
* Current consumption of soy isoflavone supplements
* Known adverse reaction to genistein, other phytoestrogens, or soy products
* Pregnant
* Unintentional weight loss of more than 10 pounds within the year
* Major or unstable medical condition
* Use of an investigational drug in the previous 30 days

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2006-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis J Smith, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with asthma were recruited from Northwestern's medical clinics and by advertisements in the community.
Pre-assignment Details: Patients with asthma were included in the study if they had mild-to-moderate disease not fully controlled on their current treatment.
Groups:
- Soy Isoflavone Supplement: This is a single blind study in which each participant was evaluated at baseline and then after receiving 100 mg of Novasoy once daily for 4 weeks.
Period: Overall Study
Arm/Group | Soy Isoflavone Supplement
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Soy Isoflavone Supplement
Number analyzed (Participants) | 13
Age Categorical [Number; unit: participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.7 (12.1)
Gender [Number; unit: participants]
  Female | 7
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Exhaled Nitric Oxide
Description: Exhaled nitric oxide at baseline (week 0) and at 4 weeks
Time Frame: 0 and 4 weeks
Population: Per protocol
Measure: Mean (Standard Deviation); unit: parts per billion (ppb)
Arm/Group | Soy Isoflavone Supplement
Number analyzed (Participants) | 13
parts per billion (ppb)
  Baseline | 67.0 (54.6)
  4 weeks | 54.8 (49.2)
Statistical Analysis 1: Comparison: Soy Isoflavone Supplement; The two groups tested were "baseline" and after "4 weeks" of treatment with the soy isoflavone supplement; Test type: Superiority or Other; p < 0.03, t-test, 2 sided

2. Secondary Outcome: Eosinophil LTC4 Synthesis
Description: Peripheral blood eosinophils were isolated before and after treatment with Novasoy, stimulated with calcium ionophore, and the amount of leukotriene C4 (LTC4) produced was measured by EIA.
Time Frame: 0 and 4 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Soy Isoflavone Supplement
Number analyzed (Participants) | 13
ng/ml
  Baseline | 3.11 (1.63)
  4 weeks | 2.07 (1.17)
Statistical Analysis 1: Comparison: Soy Isoflavone Supplement; The two groups tested were "baseline" and after "4 weeks" of treatment with the soy isoflavone supplement; Test type: Superiority or Other; p = 0.02, t-test, 2 sided

3. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1)
Description: Forced expiratory volume in one second (FEV1) measured as liters/second
Time Frame: 0 and 4 weeks
Measure: Mean (Standard Deviation); unit: liters/sec
Arm/Group | Soy Isoflavone Supplement
Number analyzed (Participants) | 13
liters/sec
  Baseline | 2.59 (0.77)
  4 weeks | 2.56 (0.92)
Statistical Analysis 1: Comparison: Soy Isoflavone Supplement; The two groups tested were "baseline" and after "4 weeks" of treatment with the soy isoflavone supplement; Test type: Superiority or Other; p = 0.88, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Duration of study = 4 weeks
Arm/Group | Soy Isoflavone Supplement
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes